CLINICAL TRIAL: NCT02357693
Title: Effect of the Association of Neurokinin-1 Receptor Antagonist Aprepitant to Dexamethasone/Ondansetron in the Incidence of Postoperative Nausea and Vomiting in High Risk Apfel Score Patients
Brief Title: Neurokinin Receptor Antagonist Associated to Ondansetron in PONV
Acronym: PONV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEP 280/12
Record Dates: First submitted 2015-01-31; First posted 2015-02-06 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: nausea, postoperative; postoperative nausea; postoperative vomiting; vomiting, postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aprepitant (Experimental): aprepitant 80 mg one hour before surgery
  Interventions: Drug: Aprepitant
- placebo (Placebo Comparator): oral placebo one hour before surgery
  Interventions: Drug: Aprepitant

INTERVENTIONS:
Drug: Aprepitant — Aprepitant or placebo will be administered to the patient before surgery
  Other Names: Emend

SUMMARY:
The purpose of this study is to determine whether patients at high risk for postoperative nausea and vomiting can benefit from aprepitant, ondansetron and dexamethasone in the perioperative period.

DETAILED DESCRIPTION:
High risk surgical patients for PONV, scheduled for laparoscopic surgery will be distributed in two groups: Group I will receive aprepitant 80 mg per os and Group II will receive placebo per os, one hour before surgery. In the operating room, patients will be submitted to combined intravenous general anesthesia plus spinal anesthesia. All patients will receive dexamethasone 4 mg and ondansetron 4 mg intravenously during the surgical procedure. After surgery, patients will be monitored for pain, nausea and vomiting during 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* high risk patients for nausea and vomiting

Exclusion Criteria:

* cardiovascular disease, or hypersensibility to any of the drugs involved in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Incidence of nausea and vomiting in postoperative period | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hazem a Ashmawi, phD, Study Director — University of Sao Paulo
Locations (1):
- Angela Maria Sousa, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Kawano H, Matsumoto T, Hamaguchi E, Manabe S, Nakagawa M, Yamada A, Fujimoto M, Tada F. Antiemetic efficacy of combined aprepitant and dexamethasone in patients at high-risk of postoperative nausea and vomiting from epidural fentanyl analgesia. Minerva Anestesiol. 2015 Apr;81(4):362-8. Epub 2014 Sep 15. PMID 25220550